CLINICAL TRIAL: NCT01584856
Title: Small Dense Low-density Lipoprotein in Patients With Prediabetes and Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-1267
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Prediabetes / Type 2 Diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
It is known that small dense LDL particles are associated with an increased cardiovascular risk. LDL particles can be separated by gradient gel electrophoresis (GGE) according to their size. The risk to suffer from coronary heart disease is 3-7 fold elevated in subjects with small dense LDL particles compared to subjects with large LDL particles. This study aims at evaluating the predictive value of small dense LDL particles in patients with prediabetes and type 2 diabetes mellitus concerning future changes in intima media thickness, flow-mediated dilation and other risk factors of atherosclerosis (e.g. insulin resistance). 60 patients with prediabetes or type 2 diabetes will be recruited for the study. Assessment will include medical history (risk factors), physical examination (blood pressure, BMI, waist-to-hip ratio), collection of serum, oral glucose tolerance test, measurement of intima media thickness and endothelial dysfunction by ultrasound. All measurements will be repeated after 2 years. Data will be analysed to assess whether the amount of small dense LDL particles can predict further structural and functional changes of the cardiovascular system or changes in the severity of the disease (insulin resistance).

ELIGIBILITY:
Inclusion criteria: - male gender

* impaired fasting glucose OR type 2 diabetes (ADA criteria)
* BMI > 25 kg/m2
* given informed consent

Exclusion criteria: - HbA1c > 9.0%

* insulin therapy
* fasting glucose > 11mmol/l
* total cholesterol > 6.5 mmol/l OR triglycerides > 2.5 mmol/l
* malignant or severe renal, hepatic, pulmonary, neurological or psychiatric disease
* alcohol or drug abuse
* HIV infection.

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prediabetes / Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kaspar Berneis, Prof. MD, Principal Investigator — University Hospital Zurich, Endocrinology and Diabetology
Locations (1):
- University Hospital Zurich, Endocrinology and Diabetology, Zurich, Canton of Zurich, Switzerland